CLINICAL TRIAL: NCT05039229
Title: Effects of Interventions to Prevent Work-related Asthma, Allergy and Other Hypersensitivity Reactions in Norwegian Salmon Industry Workers (SHInE)
Brief Title: Measures for Bioaerosol Reduction in the Salmon Industry
Acronym: SHInE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: The Research Council of Norway (Other); UiT The Arctic University of Norway (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 131052/13118
Record Dates: First submitted 2021-09-06; First posted 2021-09-09 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Asthma, Occupational; Hypersensitivity
MeSH Terms: conditions — Asthma, Occupational; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nozzles (NZ) (Experimental): Intervention with the aim of reducing bioaerosol exposure for the employees, targeting alteration of nozzles or nozzle function along the production line.
  Interventions: Other: Nozzles (NZ)
- Cleaning of surfaces (CS) (Experimental): Intervention with the aim of reducing bioaerosol exposure for the employees while cleaning their personal operating areas (work benches and part of production lines) during work operations or while cleaning floor areas.
  Interventions: Other: Cleaning of surfaces (CS)
- Control (CTR) (No Intervention): Work is to be carried out as usual without any intervention measures. Follow-up according to the same schedule as for the other intervention groups.

INTERVENTIONS:
Other: Nozzles (NZ) — Technical intervention targeting alteration of nozzles or nozzle function along the production line, e.g. by manipulation of nozzle dimensions, alteration of operating pressure or shielding of the nozzle's output stream. How the intervention is to be carried out in detail in the respective factory is to be developed in collaboration with the factory staff. This can include local specific characteristics, specific location of intervention or others.
  Arms: Nozzles (NZ)
Other: Cleaning of surfaces (CS) — Behavioural or technical intervention. This can include increased use of swabbing instead of flushing with water hoses or alterations in use of water hoses for cleaning. Examples for the latter are a reduced flushing frequency, reduction of number of employees executing the work, alterations of hose dimension or nozzles on hoses. How the intervention is to be carried out in detail in the respective factory is to be developed in collaboration with the factory staff. This can include local specific characteristics, specific location of intervention or others.
  Arms: Cleaning of surfaces (CS)

SUMMARY:
Workers in the salmon industry are at risk of developing allergies and respiratory diseases, including asthma, due to occupational exposure to bioaerosols, i.e. biological agents such as allergens, enzymes and endotoxins, in their work environment. The overall objective of this intervention trial is to identify effective and feasible control measures (interventions) that reduce exposure to these bioaerosols.

The project comprises nine salmon processing factories in northern, central and western Norway. The factories are allocated to either one of the two intervention arms or the control group. In all factories, an assessment of exposure to bioaerosols will be performed. In addition, employees will be invited to undergo a health examination and fill out a self-administered questionnaire including information on demographics, work tasks, health and health promoting factors.

The intervention trial is part of a broader study that comprises several substudies including the identification of clinically relevant allergens, investigation of exposure-response relationship between the exposure to individual bioactive agents in bioaerosols and investigations of prevalence of airway symptoms, altered lung function, skin symptoms or immunological responses indicating hypersensitivity. Finally the project includes the identification of health promoting factors that are present in the salmon processing industry.

The project is an interdisciplinary multi-center study that places great emphasis on a close dialogue between the researchers and industry in all phases of the project.

DETAILED DESCRIPTION:
The intervention trial is part of a broader study on assessment of exposure and health of workers in the salmon industry. Measurements of exposure, health examinations and questionnaire data serve as a basis for both intervention- and other substudies.

The intervention trial itself is a parallel group, three-arm non-randomized superiority trial with a 1:1:1 allocation.

Processing of salmon includes two main processes: 1) in the slaughtering department, the fish are slaughtered, sorted, automatically or manually gutted, and washed before further processing; and 2) in the filleting department, the salmon is filleted and skinned by machines before manual trimming of the fillets. The main source of exposure to fish proteins is by inhalation of wet bioaerosols containing a heterogeneous mixture of proteins, enzymes, endotoxins and microorganisms.

It is hypothesized that a reduction in exposure will cause a decrease in the prevalence of symptoms from the airways and skin, as well as sensitization, in workers of factories that implement the exposure-reducing measures.Hence, the overall aim of identifying effective and feasible control measures (interventions) that reduce exposure to these bioaerosols is to lower the risk of, or preferably prevent, the development or chronification of respiratory diseases, eczema and allergy among salmon processing workers.

The main hypothesis behind the interventions is that control measures that aim at using less water, at reduction of bioaerosol generation or at shielding workers from the production line have the potential to reduce bioaerosol exposure. The three arms of the trial are therefore 1) technical intervention targeting alteration of nozzles or nozzle function along the production line (NZ), 2) behavioral or technical intervention related to cleaning of surfaces (CS), or 3) no intervention (control). Each of the intervention arms represents a general intervention category in which details for the actual intervention are to be developed in collaboration with the factory staff to maximize the effect of the interventions.

The intervention arms NZ and CS imply measures that have the potential to reduce bioaerosol exposure for the employees, while factories in the CTR arm will not receive any active intervention measures. NZ targets alteration of nozzles or nozzle function along the production line, e.g. by manipulation of nozzle dimensions, alteration of operating pressure or shielding of the nozzle's output stream. CS focuses on reduction of bioaerosol exposure for the employees while cleaning their personal operating areas during working operations or while cleaning floor areas . This can include increased use of swabbing instead of flushing with water hoses or alterations in use of water hoses for cleaning. Examples for the latter are a reduced flushing frequency, reduction of number of employees executing the work, alterations of hose dimension or nozzles on hoses. Suggestions from employees regarding details of the intervention will be taken into account for the final design of the intervention. This can include local specific characteristics, specific location of intervention or others.

Randomization of intervention arms is not feasible due to different premises of factory infrastructure. The nine participating factories (three from each geographical region) will therefore be allocated to the study arms by the project group, reassuring that each region will cover all three study arms.

Data assessment will be done by questionnaires, exposure measurements and health examinations before (T1) and after the intervention period (T2). Interventions will start 5-8 weeks after T1, permitting technical adjustments where necessary. Interventions are to be continued until follow-up measurements at T2, 12 months after T1. Two phone calls and one physical visit are to be carried out during the intervention period.

Questionnaire data relevant for the intervention trial include background demographics, questions relevant for exposure assessment (work tasks, department, etc), as well as questions on symptoms from the eyes, the respiratory system and skin.

Health examinations will include spirometry (lung function), skin prick testing (allergic sensitization) and blood sampling (sensitization, inflammation). Exposure assessment will be done by personal exposure measurements collected in the breathing zone of workers, as well as by stationary sampling.

While all workers (approx. 1500-2000 subjects), will be eligible for answering the questionnaires, the number of invitees for health examination and exposure assessments will be much lower (ca 900 and 216, respectively), due to logistical and timely constraints.

Sample size calculations was performed for the primary outcome; the effect of interventions in reducing the concentration of bioaerosols (total protein) in salmon processing plants. The inclusion of 24 workers with 2 repeated measurements in each of the three intervention arms (see section on inclusion criteria above) will give a total of 432 measurements (144 measurements in each of the intervention arms). According to the sample size calculations, 133 exposure measurements of total proteins in each of the intervention arms give a power of 80% of detecting a 20% reduction of exposure (significance level of 0.05). The corresponding number of measurements needed to detect a reduction in exposure of 40 and 30% were 34 and 59 measurements, respectively. Hence, 144 measurements as aimed at in the present study will ensure a buffer of about 8% in order to account for rejection of measurements due to sampling errors. The number of exposure measurements per work shift will also be limited by logistical constraints.

ELIGIBILITY:
Eligibility criteria will differ depending on the type of data gathering volunteers participate in:

1. Questionnaire Inclusion Criteria: All workers employed in the factory Exclusion Criteria: No restrictions
2. Exposure assessment study

   Inclusion Criteria: Participants (12 workers each day, two repeated measurements = 24 workers) will be collected at random among workers having the following work stations/tasks during the study period:

   Monday and Thursday (n=12 workers): Slaughtering department (n=5), filleting department (n=4) and other (n=3).

   Tuesday and Wednesday (n=12 workers): Slaughtering department (n=3), filleting department (n=3), packing department (n=2), laboratory/technical department (n=2) and central control room/administration (n=2).

   Exclusion Criteria: Not working in those areas, not able to wear backpack with equipment.
3. Cross-week follow-up (Monday to Thursday) Inclusion Criteria: Participant in both 1 and 2, i.e. having filled out questionnaire and participated in exposure measurement on mondays.

   Exclusion Criteria: Not fulfilling inclusion criteria, not able to wear backpack with equipment.
4. Health examinations Inclusion criteria: All subjects working in the factories during the field work period of four days will be eligible. However, due to logistic constraints we aim to invite at least 20 subjects each day, primarily those working in the salmon production line. Those invited will be randomly selected according to a distribution between slaughtering, filleting and others (ratio 5:4:3).

Exclusion criteria:

* For spirometry measurements: heart attack, operation on eyes, stomach or in the chest region in the course of the last three months, ongoing treatment for tuberculosis or other respiratory infection, pregnancy
* For skin prick tests: pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of salmon processing workers' personal exposure to inhalable protein | Measurements at T1 compared to T2, 12 months after T1.
  Change in inhalable total protein (ug/m3) in the workers' breathing zone from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences in mean concentration of full shift measurements (8 hours) between intervention groups and between intervention groups and control group will be analyzed.

SECONDARY OUTCOMES:
Change of salmon processing workers' personal exposure to proteases | Measurements at T1 compared to T2, 12 months after T1.
  Change in concentration of proteases (ng/m3) in the workers' breathing zone from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences in mean concentration of full shift measurements (8 hours) between intervention groups and between intervention groups and control group will be analyzed.
Change in area concentration of airborne total protein (stationary measurements) | Measurements at T1 compared to T2, 12 months after T1.
  Change in total protein (ug/m3, inhalable aerosol fraction) from stationary measurements in relevant areas of the salmon production line from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences in mean concentration of full shift measurements (8 hours) between intervention groups and between intervention groups and control group will be analyzed.
Change of salmon processing workers' personal exposure to airborne fish allergens | Measurements at T1 compared to T2, 12 months after T1.
  Change in concentration of total aerosol fraction of fish allergens (ng/m3) in the workers' breathing zone from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences in mean concentration of full shift measurements (8 hours) between intervention groups and between intervention groups and control group will be analyzed.
Change of salmon processing workers' personal exposure to airborne endotoxins | Measurements at T1 compared to T2, 12 months after T1.
  Change in mean concentration of inhalable total endotoxin units (EU/m3) in the workers' breathing zone from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences in mean concentration of full shift measurements (8 hours) between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' self-reported symptoms from the upper airways | Data collected at T1 compared to T2, 12 months after T1.
  Since the investigators expect to have a significant "loss to follow-up" from T1 to T2,the investigators will analyze change in prevalence of self-reported symptoms from the nose from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Prevalence of symptoms from the respiratory system will be assessed using information reported by participants through a questionnaire that includes standardized questions on respiratory symptoms (upper and lower airways), allergic status and malaise (European Community Respiratory Health Survey, ECRHS). Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' self-reported symptoms from the lower airways | Data collected at T1 compared to T2, 12 months after T1.
  Since the investigators expect to have a significant "loss to follow-up" from T1 to T2, the investigators will analyze change in prevalence of self-reported symptoms from the chest from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Prevalence of symptoms from the respiratory system, as well as the asthma symptom score (0-5) will be assessed using information reported by participants through a questionnaire that includes standardized questions on respiratory symptoms (upper and lower airways), allergic status and malaise (European Community Respiratory Health Survey, ECRHS). Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' self-reported eye symptoms | Data collected at T1 compared to T2, 12 months after T1.
  Since the investigators expect to have a significant "loss to follow-up" from T1 to T2, the investigators will analyze change in prevalence of self-reported symptoms from the eye pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Prevalence of eye symptoms will be assessed using information reported by participants through the a set of standardized questions in a questionnaire.Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' lung function at group level (FEV1 in % of predicted) | Measurements at T1 compared to T2, 12 months after T1.
  Change in proportion of participants having a decline in maximum forced expired volume in 1 second (FEV1 in % of predicted), from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' lung function at individual level (maximum forced expired volume in 1 second (FEV1)/forced vital capacity (FVC) ratio) | Data collected at T1 compared to T2, 12 months after T1.
  Mean of individual change in maximum forced expired volume in 1 second (FEV1) in % of forced vital capacity (FEV1/FVC ratio), from pre-intervention (baseline, T1) to post-intervention (follow-up, T2) for individuals, provided low loss-to follow up. Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' cross-shift lung function (FEV1) | Measurements at T1 compared to T2, 12 months after T1.
  Change in mean difference between pre-shift values and post-shift values (cross-shift) in maximum forced expired volume in 1 second (FEV1, in liter and % of predicted) of individual salmon processing workers from pre-intervention (baseline, T1) to post-intervention (follow-up, T2) .Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' cross-week lung function (FEV1) | Measurements at T1 compared to T2, 12 months after T1.
  Change in mean difference between pre-shift values on Monday and post-shift values on Thursday (cross-week) in maximum forced expired volume in 1 second (FEV1, in liter and % of predicted) of individual salmon processing workers from pre-intervention (baseline, T1) to post-intervention (follow-up, T2) .Differences between intervention groups and between intervention groups and control group will be analyzed.
Incidence of salmon processing workers' sensitization to salmon | Measurements at T1 compared to T2, 12 months after T1.
  Registration of number of salmon workers that are newly sensitized to salmon at follow-up. Sensitization will be assessed by serum immunoglobulin E (IgE) specific to salmon proteins. Individuals that are negative for specific immunoglobulin E (IgE) at pre-intervention (baseline, T1) and positive at post-intervention (follow-up (T2) will be registered as an incidence case. Differences between intervention groups and between intervention groups and control group will be analyzed.
Change in salmon processing workers' self-reported skin symptoms | Data collected at T1 compared to T2, 12 months after T1.
  Since the investigators expect to have a significant "loss to follow-up" from T1 to T2, the investigators will analyze change in prevalence of self-reported skin symptoms from pre-intervention (baseline, T1) to post-intervention (follow-up, T2). Skin symptoms will be assessed using information from a questionnaire that includes standardized questions on eczema, other symptoms from the skin and urticaria (Nordic Occupational Skin Questionnaire, The Nordic Occupational Skin Questionnaire NOSQ-2002). Differences between intervention groups and between intervention groups and control group will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Berit E Bang, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of Nothern Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD)-sharing will be restricted due to sensitive health data. Where possible, de-identified data will be made available after the end of the project period for researchers whose aim is to increase knowledge in the field of allergy, hypersensitivity and/or occupational health. A data handling group comprising at least one representative from each location will consider written applications from external researchers before possibly releasing individual data. More details regarding criteria for applications and which data will be made available is under preparation.

REFERENCES:
- [Background] Hoper AC, Kirkeleit J, Thomassen MR, Irgens-Hansen K, Hollund BE, Fagernaes CF, Svedahl SR, Eriksen TE, Grgic M, Bang BE. Effects of Interventions to Prevent Work-Related Asthma, Allergy, and Other Hypersensitivity Reactions in Norwegian Salmon Industry Workers (SHInE): Protocol for a Pragmatic Allocated Intervention Trial and Related Substudies. JMIR Res Protoc. 2023 Jul 19;12:e48790. doi: 10.2196/48790. PMID 37467018